CLINICAL TRIAL: NCT04555395
Title: The Differences Between Gonadal and Extra-gonadal Malignant Teratomas in Both Genders and the Effects of Chemotherapy
Brief Title: The Differences Between Gonadal and Extra-gonadal Malignant Teratomas
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Shanghai 10th People's Hospital, Shanghai 10th People's Hospital
Other Study IDs: malignant teratomas
Record Dates: First submitted 2020-09-15; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: SEER Database
MeSH Terms: interventions — Survival Rate

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- gonadal
  Interventions: Other: survival rates
- extra-gonadal
  Interventions: Other: survival rates
- chemotherapy
  Interventions: Other: survival rates
- without chemotherapy
  Interventions: Other: survival rates

INTERVENTIONS:
Other: survival rates — survival rates

SUMMARY:
A tumor comprising of different types of tissues (such as hair, muscle, bone, etc.) is known as a teratoma. It is a type of germ cell (cells that make sperm or eggs) tumor. When these germ cells have rapid cancerous growth, then such a teratoma is called a malignant teratoma. We have studied the differences between gonadal and extra-gonadal malignant teratomas and the effects of chemotherapy in both genders.

Methods: The samples of 3799 male and 1832 female patients with malignant teratoma samples, between the ages of 1 and 85+ years, were selected from the years 1973 to 2014. Trends in incidence, estimated prevalence, incidence rates, and frequency were calculated in gonadal and extra-gonadal tumors with age adjustment. The fiveyear observed, expected, and relative survival rates were analyzed to study the prognosis.

ELIGIBILITY:
The registry used in our study was the SEER 9 registries Custom Data (with additional treatment fields), Nov 2016 Submission (1973-2014) < Katrina/Rita Population Adjustment> - Linked to County Attributes -Total United States, 1969-2015 Counties, National Cancer Institute, DCCPS (Division of Cancer Control and Population Sciences), Surveillance Research Program, released April 2017, based on the November 2016 submission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry used in our study was the SEER 9 registries Custom Data (with additional treatment fields), Nov 2016 Submission (1973-2014) < Katrina/Rita Population Adjustment> - Linked to County Attributes -Total United States, 1969-2015 Counties, National Cancer Institute, DCCPS (Division of Cancer Control and Population Sciences), Surveillance Research Program, released April 2017, based on the November 2016 submission.
Sampling Method: Probability Sample
Enrollment: 3799 (Actual)
Dates: Start 1973-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
survival rates | 1973-2014